CLINICAL TRIAL: NCT06295237
Title: Comparison of the Prevalence of Asynchronies During Mechanical Ventilation With Manual Versus Automatic Adjustment Ventilator Settings Using the INTELLISYNC+® (HAMILTON) Tool. A Randomized Controlled Study
Brief Title: Automatic Adjustment for Asynchronies During Mechanical Ventilation
Acronym: i-Sync
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility. Intermediate analysis shows no difference in outcome variables
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Principal Investigator, Miguel Sanchez Garcia, Director Critical Care Department, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: i-Sync
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Mechanical Ventilation Complication
Keywords: Asyncronies; Mechanical ventilation; Automatic detection and adjustment

STUDY DESIGN:
Intervention Model Description: Two 2-hour periods: 1) "off mode" consisting of a control period with optimized ventilator parameters and 2) "on mode" with an active automated detection and adjustment for asynchronies. The starting first period is randomized.
Who Masked: Outcomes Assessor
Masking Description: Anonymized evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (No Intervention): Optimized ventilator settings to control and reduce the number of asynchronies
- Activated automatic detection and adjustment of asynchronies (Active Comparator): Active mode of a mechanical ventilator software automatically detecting and adjusting ventilator parameters to control or reduce the number of events.
  Interventions: Device: Intellisync+

INTERVENTIONS:
Device: Intellisync+ — mechanical ventilator software automatically detecting and adjusting ventilator parameters to control or reduce the number of events.
  Arms: Activated automatic detection and adjustment of asynchronies

SUMMARY:
Asynchronies between the patient and the artificial ventilator are a frequent problem. They may cause altered sleep, ventilator-induced lung injury, prolong length of ICU stay, cause neuro-psycologic complications and increase mortality. Although reducing their incidence through ventilator setting adjustments is possible, they frequently go undetected and it also requires that attendings remain at the bedside to repeatedly modify ventilator parameters. Ventilator systems may detect and automatically adjust parameters of mechanical ventilation. This would avoid delays in detection and adjustment if the intensivist is not immediately available. The investigators intend to study an automatic detection and adjustment tool which is incorporated in the ventilator software.

DETAILED DESCRIPTION:
The prevalence and time course of asynchronies will be evaluated in subjects under invasive (n=40) or non-invasive (n=40) mechanical ventilation. Intensivist-optimized ventilator settings will be compared to a software tool (Hamilton ventilators, Intellisync+) in its capacity to control and adjust the triggering and cycling by analysis of the ventilator curves.

The outcome variable is the percentage of the duration of asynchronies during the two 2-hour study periods.

This pilot study has a prospective, randomized cross-over design. The order of the 2 study periods will be randomized to either start with "control" with manual adjustment or "automated adjustment" with Intellisync+.

The total sample size is 80 subjects, 40 receiving invasive mechanical ventilation and 40 on non-invasive mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Age >17 years
* Partial ventilatory support ("SPONT" mode) connected to Hamilton C1 model, irrespective of chronic restrictive or obstructive lung disease, categorized by RCexp (Expiratory time constant): restrictive (RCExp <0.6); obstructive (RCExp >0.9); normal (RCExp 0.6 - 0.9).
* Software version SW3.0.0 or superior and the IntelliSync+ software tool available in invasive and non-invasive ventilation.
* Presence of asyncronies in pressure and volume curves tracings of the ventilator.
* Signed informed content.

Exclusion Criteria:

* Pregnant
* On extracorporeal respiratory support (ECMO or ECCO2R)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Duration of asyncronies | two hours per study arm
  duration of asyncronies expressed as percentage of time during the respective 2-hour study periods

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Sanchez-Garcia, MD, Study Chair — Hospial Clinico San Carlos
Locations (1):
- Hospital Clinico San Carlos, Madrid, Madrid, Spain